CLINICAL TRIAL: NCT04304833
Title: Innovative Care of Older Adults With Chronic Heart Failure (I-COACH): A Comparative Effectiveness Clinical Trial
Brief Title: Innovative Care of Older Adults With Chronic Heart Failure: A Comparative Effectiveness Clinical Trial (I-COACH)
Acronym: I-COACH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in PI
Sponsor: University of Arkansas (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 260092
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The provider-directed management model is the current care standard for patients with HF; care delivery consists of office and emergency visits, with telephone or in person communications. The mHealth care management model consists of real time bio-monitoring kits and telemedicine visits using a secure wireless gateway with a cloud-based clinician portal connected to a Bluetooth-paired Android Tablet. Daily readings are transmitted to a 24-hour RN call center and triaged per protocols.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Provider-Based Care Model Arm (Active Comparator): Non-connected home vital sign equipment will be given to patients in this group. The patients in the group will be instructed to record their daily readings on a paper log provided by the research team. These monitoring devices will not transmit readings to a centralized location and no one will be alerted to out-of-range readings or compliance with taking daily vital sign measures. At the front page of the log, normal ranges will be described with brief instructions about what participants/caregivers should do if their readings are out-of-range. Logs will be collected at baseline, 3-months and 6-months.
  Interventions: Other: Provider-Based Care Model Arm
- mHealth Model Arm (Experimental): Connected home vital sign equipment (mHealth) will be given to patients in this group. The patients will be instructed to take their daily readings, which will automatically be sent to the secure cloud-based software. If the readings are out-of-range, the Registered Nurse (RN) Call Center will be automatically alerted and the event will be triaged. Daily measures and medical follow-up from the measures will be counted and collected at baseline, 3-months, and 6-months.
  Interventions: Behavioral: mHealth Model Arm

INTERVENTIONS:
Other: Provider-Based Care Model Arm — The PI will be supplementing standard care by providing and training each patient in the use of an analog (not internet connected) vital sign kit for 6 months: weight scale, blood pressure cuff, pulse oximeter. A Log for recording their vital sign measures.
  Arms: Provider-Based Care Model Arm
Behavioral: mHealth Model Arm — The PI will provide each patient with weight scale, blood pressure cuff, & pulse oximeter kit connected to a Bluetooth-paired Android Health Tablet for 6 months. Daily vital sign readings will be sent to the secure cloud-based software. If the readings are out-of-range, the Registered Nurse Call Center will be automatically alerted and triaged.
  Arms: mHealth Model Arm

SUMMARY:
An estimated 6.5 million adults in the U.S. have Heart Failure (HF) and the prevalence is increasing. HF is characterized by poor quality of life but this is amenable to self-management. However, the amount of support available from providers to help manage complications is far beyond what is feasible. The complex needs of these patients require a new vision for delivery of health care services, such as an mHealth management model. mHealth technologies such as blue-tooth enabled BP, heart rate, weight, and pulse oximetry remote monitoring permit sharing of immediate biometric data and video messages with providers and instantaneous feedback to patients before symptom crises, that is, when and where patients need it.

DETAILED DESCRIPTION:
An estimated 6.5 million adults in the U.S. have Heart Failure (HF) and the prevalence is increasing. HF is characterized by poor quality of life but this is amenable to self-management. However, the amount of support available from providers to help manage complications is far beyond what is feasible. The complex needs of these patients require a new vision for delivery of health care services, such as an mHealth management model. mHealth technologies such as blue-tooth enabled BP, heart rate, weight, and pulse oximetry remote monitoring permit sharing of immediate biometric data and video messages with providers and instantaneous feedback to patients before symptom crises, that is, when and where patients need it.

This is a single-blinded comparative effectiveness randomized controlled trial conducted in a real-world setting. A sample of 400 dyads, that is older patients with HF (>55 years) and their caregivers, will be recruited from a large medical center and randomly assigned to one of two arms: 200 dyads to a provider-directed model or 200 dyads to the mHealth management model. The provider-directed management model is the current care standard for patients with HF; care delivery consists of office and emergency visits, with telephone or in person communications. The standard of care will be augmented by providing home equipment kits with weight scale, blood pressure, pulse oximetry devices and a Log to record data. The mHealth care management model consists of real time bio-monitoring kits and telemedicine visits using a secure wireless gateway with a cloud-based clinician portal connected to a Bluetooth-paired Android Tablet. Daily readings are transmitted to a 24-hour RN call center and triaged per protocols. Outcomes informed a prior by community stakeholders to be most important at the patient, caregiver, and health systems-levels will be collected and compared at baseline, 3- and 6- months: 1) For the patient: self-care of HF; confidence and self-efficacy to manage care, symptoms, medications and treatments; HF knowledge; mental and physical health, health distress, informational support, equipment usability, and quality of life. 2) For the caregiver: caregiver burden and health. 3) For the Health System: patient satisfaction, hospital, emergency & provider visits, and mortality. Differential benefits for subsets of participants will be evaluated according to patient characteristics (socio-demographical, rurality, etc.). Evaluation of mediation variables will enhance our understanding of underlying processes. This research has the potential to revolutionize care for high-cost and high-need patients such as those with HF.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 55 years with HF (documented in medical record).
* Has capacity to understand informed consent.
* Able to stand (briefly) without assistance.
* Has a designated caregiver.
* Agrees to be followed (treated) by UAMS physician/provider for 6 months after discharge.

Exclusion Criteria:

* Speaks a language other than English or Spanish.
* Active psychosis or other severe cognitive disorder that interferes with capacity to understand and comply with study procedures.
* A history of drug or alcohol abuse in the past 90 days (documented in medical record).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Weber, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Rhoads SJ, McSweeney J, Sadaka H, Jin J, Pirtle C, Sanford J. Experiences of Older Adults with Heart Failure Using Telemedicine During the COVID-19 Pandemic: A Qualitative Study. Telemed J E Health. 2025 Feb;31(2):191-199. doi: 10.1089/tmj.2024.0005. Epub 2024 Sep 30. PMID 39348299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled and assessed in the study are HF patients. Caregivers were not enrolled.
Period: Overall Study
Arm/Group | Provider-Based Care Model Arm | mHealth Model Arm
Started (Participants enrolled and assessed in the study are HF patients. Caregivers were not enrolled.) | 12 | 14
Completed | 8 | 12
Not Completed | 4 | 2
Not completed — Due to the pandemic in person visits were not allowed | 4 | 2

BASELINE CHARACTERISTICS:
Population: Participants enrolled and assessed in the study are HF patients. Caregivers were not enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Provider-Based Care Model Arm | mHealth Model Arm | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (6.48) | 64.67 (8.89) | 63.60 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We had participants withdraw from the study.
  Participants
    number analyzed (Participants) | 4 | 6 | 10
    Female | 3 | 1 | 4
    Male | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the COVID-19 pandemic our study was drastically impacted and our participant pool was decreased.
  Participants
    number analyzed (Participants) | 4 | 6 | 10
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 4 | 6
    White | 2 | 2 | 4
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Self-Care of Heart Failure Maintenance Scale (SCHFI)
Description: self care scores on a scale range from 70 to 100, mean (SD). The SCHFI uses a Likert-type scale, with responses ranging from 1 (never) to 5 (always). The SCHFI also includes scales for self-care management and self-care confidence. Higher scores on the SCHFI indicate better self-care. A score of less than 70 on any of the subscales is considered inadequate self-care.
Time Frame: Change from Baseline, 3 months, and 6 months
Population: The study was terminated by mutual agreement by the funding agency and UAMS due to circumstances of the pandemic which made it impossible to recruit patients in the hospital and their caregivers were not allowed in the hospital setting.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider-Based Care Model Arm | mHealth Model Arm
Number analyzed (Participants) | 8 | 12
score on a scale
  Baseline | 75.50 (14.55) | 83.67 (13.41)
  3 Month | 80.00 (8.72) | 99 (1.41)
  6 Month | 83.50 (3.42) | 74.67 (21.39)

2. Secondary Outcome: Promis 43v2.1 Health Profile Anxiety 6a
Description: subscale of questionnaire that measures anxiety. Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population. Min/max range is 39.1-82.7
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Promis 43v2.1 Health Profile Depression 6a
Description: subscale of questionnaire that measures depression. Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population. Min/Max range 38.4-80.3
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Promis 43v2.1 Health Profile Fatigue 6a
Description: subscale of questionnaire that measures fatigue. Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population. Min/Max range 33.4-76.8
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Promis 43v2.1 Health Profile Pain Interference 6a
Description: subscale of questionnaire that measures pain. Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population. Min/Max range 41.1-76.3
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Promis 43v2.1 Health Profile Physical Function 6b
Description: subscale of questionnaire that measures physical function. Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population. Min/Max range 21.6-58.7
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Promis 43v2.1 Health Profile Sleep Disturbance 6a
Description: subscale of questionnaire that measures sleep disturbance. Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population Min/Max Range 31.7-76.1
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Promis 43v2.1 Health Profile Ability to Participate in Social Roles and Activities 6a
Description: subscale of questionnaire that measures the ability to participate in social roles and activities . Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population. Min/Max Range 26.7-65
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Promis 43v2.1 Health Profile PROMIS Pain Intensity Item (Global07)
Description: subscale of questionnaire that measures pain intensite. Scoring for this PROMIS instrument uses Item Response Theory (IRT), a family of statistical models that link individual items to a presumed underlying trait or concept represented by all items in the item bank. Score of 50 on any domain is the average. Greater than 50 likely represents somewhat sicker people than the general population. Min/Max range 0-10
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

10. Secondary Outcome: Medical Outcomes Study MOS Health Distress Scale
Description: questionnaire assesses psychological impact/health distress
Time Frame: Change from Baseline, 3 months, and 6 months
Reporting Status: Not Posted

11. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire (MLHFQ)
Description: questionnaire to assess quality of life. Scoring for the MLHFQ ranges from 0 to 105, the higher the score the more affected, over the past 4 months, the individual is by their heart failure.
Time Frame: Change from Baseline to 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Zarit Caregiver Burden Scale
Description: questionnaire to Assess caregiver perception of burden. Scoring of the Zarit Burden Interview ranges from 0-88, the higher the score, the more severe the burden on the caregiver.
Time Frame: Change from baseline to 6 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Optum SF36v2 Health Survey
Description: questionnaire to Assess caregiver health
Time Frame: Change from baseline to 6 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: questionnaire to Assess patient's satisfaction with care received
Time Frame: Change from baseline to 3 months and 6 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Treatment Visits
Description: number of medical treatment visits
Time Frame: Change from baseline to 3 months and 6 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Mortality
Description: death
Time Frame: 3 months and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6.5 months
Description: A risk to study participants is the potential for loss of confidentiality of study data (study participants are those enrolled with CF; caregivers were not enrolled)
Arm/Group | Provider-Based Care Model Arm | mHealth Model Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

LIMITATIONS AND CAVEATS:
That the sample size was too small for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT04304833/Prot_SAP_000.pdf